CLINICAL TRIAL: NCT05776979
Title: Post-Transplant Maintenance Therapy With Isatuximab Plus Lenalidomide for High-Risk Multiple Myeloma Patients
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-0028; NCI-2023-02219 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2023-03-08; First posted 2023-03-20 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — isatuximab; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- isatuximab plus lenalidomide after an autologous stem cell transplantation (ASCT) (Experimental): Both isatuximab and lenalidomide are FDA approved and commercially available for the treatment of relapsed or refractory MM (MM that has come back or stopped responding to treatment). Participants will begin taking the study drugs about 60-180 days after your ASCT. Participants may receive the study drugs for about 3 years. After that, participants will have follow-up visits 1 time a year for the 3 years after your last dose of study drugs
  Interventions: Drug: Isatuximab; Drug: lenalidomide

INTERVENTIONS:
Drug: Isatuximab — Given by vein over about 75 minutes
  Other Names: SAR650984
Drug: lenalidomide — Given by PO

SUMMARY:
To learn if isatuximab can help to control highrisk MM when given in combination with lenalidomide after an autologous stem cell transplantation (ASCT).

DETAILED DESCRIPTION:
Objectives:

Primary Objectives

1. Compare progression-free survival at 3 years with historical control rate of 50%.

Primary endpoint

1. Progression-free survival at 3 years, measured from the date of transplant to the date of progression or death.

Secondary objectives:

1. Assess minimal residual disease (MRD) rate at 12 months after starting Isatuximab maintenance therapy
2. Assess overall best response rate (defined as the occurrence of VGPR or better and CR/sCR) before the 4th Isatuximab cycle, and at 12, 24, and 36 months after starting maintenance therapy
3. Assess MRD rate before 4th Isatuximab cycle and at 24 months after starting maintenance therapy
4. Assess duration of response (DOR)
5. Assess overall survival (OS)
6. Assess safety

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients 18 to 72 years old, with newly diagnosed symptomatic (according to the revised 2014 IMWG criteria as summarized in Appendix A) myeloma. Patients must have measurable disease at diagnosis defined by any of the following:

   * Serum M-protein ≥1 g/dL (for IgA ≥0.5 g/dL) or urine M-protein ≥200 mg/24 hours
   * For oligosecretory myeloma, involved serum free light chain (FLC) level ≥10 mg/dL, provided serum FLC ratio is abnormal
   * For non-secretory myeloma, > 1 focal lesions measurable by imaging
2. Subjects must have high-risk myeloma defined as followed:

   * R-ISS stage II or III patients (Appendix B)
   * ISS stage III (Appendix B)
   * ≥ 3 copies +1q21 in patients with ISS Stage II/III or R-ISS Stage II/III
   * Presence of del(17p) cytogenetic abnormality regardless of ISS/R-ISS Stage
   * Presence of at least 2 high-risk genetic abnormalities [del(17p), t(4;14), t(14;16), t(14;20), +1q21] regardless of ISS/R-ISS stage
3. English and non-English speaking patients are eligible.
4. Karnofsky performance score of at least 70% and/or ECOG PS ≤2
5. Underwent ASCT using a conditioning regimen consisting of single agent Melphalan or a combination of Busulfan and Melphalan with adequate cell count recovery after transplant without the need for growth factor support or transfusions within 7 days from the lab test:

   * Absolute neutrophil count (ANC) ≥1000 /µL
   * Hemoglobin ≥8 g/dL
   * Platelet count ≥50,000 /µL
6. Patients must have achieved partial response (PR) or better prior to starting maintenance therapy.
7. Adequate major organ system function as demonstrated by:

   * Serum creatinine clearance equal or more than 30 ml/min (calculated with Cockcroft- Gault formula).
   * Total bilirubin equal or less than 2.0 mg/dL (equal or less than 3.0 mg/dL for patients with Gilbert's disease).
   * ALT or AST equal or less than 3 times the upper normal for adults.
8. Patient or patient's legal representative, parent(s) or guardian should provide written Internal Review Board (IRB)-approved informed consent.
9. Female patients included must not be pregnant or lactating. Females of childbearing potential must have (before starting treatment) a negative serum or urine pregnancy test with a sensitivity of at least 25 mIU/mL within 10-14 days prior to and again within 24 hours prior to starting Isatuximab and with each cycle of study treatment. Females of childbearing potential must refrain from becoming pregnant and commit to either apply highly effective method of birth control (two reliable methods of birth control) or continue abstinence from heterosexual intercourse during study period and for at least 5 months after last dose of Isatuximab. Patients who receive Lenalidomide should continue to follow REVLIMID REMSTM requirements.
10. Men of reproductive potential must agree to follow accepted birth control methods and refrain from sperm donation for the duration of the study and for at least 5 months after last dose of Isatuximab. Patients who receive Lenalidomide should continue to follow REVLIMID REMSTM requirements.

Exclusion Criteria

1. Progression of myeloma, as defined by the IMWG criteria (Appendix C), prior to initiation of maintenance therapy
2. Patients receiving any other investigational agents within 14 days or 5 half-lives of the investigational drug prior to initiation of study intervention. Exceptions can be granted after discussing with PI.
3. History of allergic reactions attributed to compounds of similar chemical or biologic composition to any of the study drugs. Hypersensitivity or history of intolerance to steroids, mannitol, pregelatinized starch, sodium stearyl fumarate, histidine (as base and hydrochloride salt), arginine hydrochloride, poloxamer 188, sucrose or any of the other components of study intervention that are not amenable to premedication with steroids and H2 blockers or would prohibit further treatment with these agents.
4. Known hypersensitivity or desquamating rash to either thalidomide or lenalidomide.
5. Participants must not have an active infection requiring treatment.
6. Participants must not have an uncontrolled intercurrent illness including, but not limited to, an uncontrolled hypertension (systolic >170, diastolic >100 despite antihypertensive therapy), symptomatic congestive heart failure (Class III or IV as defined by the New York Heart Association (NYHA) functional classification system), acute coronary syndrome, liver cirrhosis, and/or cognitive impairments/psychiatric illness/social situations that would limit compliance with study requirements. PI is the final arbiter of this criterion.
7. Major surgery within 4 weeks before initiating study treatment.
8. HIV-positive patients and/or active hepatitis A, B or C infections.

Ages: 18 Years to 72 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Estimated)
Dates: Start 2023-08-17 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5 | through study completion; an average of 1 year.

CONTACTS AND LOCATIONS:
Overall Officials: Muzzaffar Qazilbash, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org